CLINICAL TRIAL: NCT02430038
Title: The Sono-VE Study: Assessing the Acceptability and Feasibility of Transperineal Ultrasound and Developing an Ultrasound Based Predictive Model for Labour Outcome.
Brief Title: Transperineal Ultrasound to Assess the Progress of Labour
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); KU Leuven (Other); Norwegian University of Science and Technology (Other); British Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 14HH2428
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Placenta Praevia; Vaginismus
Keywords: transperineal ultrasound; labour; sonopartogram; prediction model
MeSH Terms: conditions — Placenta Previa; Vaginismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acceptability: To assess acceptability of intervention. Some patients from this group also participated in the other groups.
- Feasibility: Is it possible for ultrasound to measure labour parameters, where vaginal examinations are best avoided e.g. vaginismus or contraindicated (PPROM) with controls. Some patients from this group also participated in the other groups.
- Predictive Model: Nulliparous term labouring women with cephalic presentation. Some patients from this group also participated in the other groups.

SUMMARY:
This is a prospective observational study of transperineal ultrasound between 24-42 weeks gestation and a prospective longitudinal observational study in all term (37-42 weeks) labouring women.

DETAILED DESCRIPTION:
This is a prospective observational study of transperineal ultrasound between 24-42 weeks gestation and a prospective longitudinal observational study in all term (37-42 weeks) labouring women.

AIMS:

This study aims to firstly assess the effectiveness and acceptability of transperineal ultrasound in women presenting between 24 and 42 weeks gestation in comparison with digital vaginal examination (VE). Secondly, in all term (37-42 weeks) labouring women, investigators aim to create an ultrasound based labour record, "a sonopartogram" and from this develop a predictive model for the outcome of labour.

ELIGIBILITY:
Inclusion Criteria:

* Gestation 24-42 completed weeks at study entry
* Aged 18-44
* Cephalic
* Singleton pregnancies
* Nulliparous
* Multiparous (excluded for the term predictive model group)
* Multiple pregnancies (excluded for the term predictive model group)
* Established (Active) phase of labour (included for the term predictive model group) o Clinician opinion that patient is in the established phase of labour according to the current NICE guidelines

Exclusion Criteria:

* Younger than 18 years.
* Imminent iatrogenic intention to deliver
* Life threatening maternal or fetal compromise needing immediate medical attention and/or delivery
* Women who in the opinion of the researcher by virtue of language or learning impairment would be unable to give fully informed consent to the study.
* Miscarriage
* Intra-uterine death
* Previous cervical surgery eg. cone biopsy, cervical cerclage. Note- Single LLETZ is not excluded.
* Non-cephalic presentations
* Multiple pregnancies (for the term predictive model group)
* Multiparous patients (for the term predictive model group)
* Not in established labour (for the term predictive model group)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1: acceptability and feasibility group
  Group 2: predictive model group
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lees, MD MRCOG, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study aimed to firstly assess the feasibilty and acceptability of transperineal ultrasound in women presenting between 24 and 42 weeks gestation in comparison with digital vaginal examination (VE). Secondly, in all term (37-42 weeks) labouring women, we aim to create an ultrasound based labour record, "a sonopartogram" and from this develop a predictive model for the outcome of labour.
Pre-assignment Details: Recruitment start date 22/04/2015 Recruitment end date 19/01/2018
Groups:
- Acceptability; Feasibility: Where vaginal examinations are best avoided e.g. vaginismus or contraindicated (PPROM) with controls
- Predictive Model: Nulliparous term labouring women with cephalic presentation
Period: Overall Study
Arm/Group | Acceptability | Feasibility | Predictive Model
Started | 119 | 195 | 270
Minimum Recruitment | 42 | 100 | 270
Completed (119 women recruited) | 119 | 195 (270 recruited) | 269
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Acceptability and Feasibilty; Feasibility: Where vaginal examinations are best avoided e.g. vaginismus or contraindicated (PPROM) with controls
- Total: Total of all reporting groups
Arm/Group | Acceptability and Feasibilty | Feasibility | Predictive Model | Total
Number analyzed (Participants) | 119 | 195 | 270 | 584
Age, Continuous [Median (Standard Deviation); unit: years] | 31.2 (5.3) | 31 (4.8) | 31.0 (5.1) | 31 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 195 | 270 | 584
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 119 | 195 | 270 | 584
  Unknown or Not Reported | 0 | 0 | 0 | 0
Regional analgesia [Count of Participants; unit: Participants] | 95 | 178 | 211 | 484

OUTCOME MEASURES:

1. Primary Outcome: Caesarean Delivery
Description: Number of Caesarean deliveries in the prediction group
Time Frame: 24 months
Population: Total number of Caesarean deliveries
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptability | Feasibility | Predictive Model
Number analyzed (Participants) | 0 | 0 | 269
Participants |  |  | 79

2. Primary Outcome: Acceptability of Intrapartum Ultrasound
Description: Acceptability of transabdominal and transperineal ultrasound to pregnant and labouring women. Use of modified W-DEQ questionnaires pre and post assessment. We recorded the number of women who completed both questionnaires.
Time Frame: 24 months
Population: Only analysing patients in the acceptability arm for this primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptability | Feasibility | Predictive Model
Number analyzed (Participants) | 119 | 0 | 0
Participants | 104 | 0 | 0

3. Primary Outcome: Feasibility of Ultrasound Labour Parameters
Description: The outcome was the number of women who had all labour parameters measured by ultrasound.
Time Frame: 24 months
Population: The outcome was the number of women who had all labour parameters measured by ultrasound.
Measure: Count of Participants; unit: Participants
Arm/Group | Acceptability | Feasibility | Predictive Model
Number analyzed (Participants) | 0 | 195 | 0
Participants | 0 | 168 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse event definition in study protocol. No adverse events reported.
Groups:
- Acceptability: To assess acceptability of intervention
- Feasibility of the Study: To assess if ultrasound can measure labour parameters where vaginal examinations are best avoided e.g. vaginismus or contraindicated (PPROM) with controls
Arm/Group | Acceptability | Feasibility of the Study | Predictive Model
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/195 | 0/270
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/195 | 0/270
Other Adverse Events (participants affected / at risk) | 0/119 | 0/195 | 0/270

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT02430038/Prot_SAP_000.pdf